CLINICAL TRIAL: NCT06433778
Title: Vonicog Alfa (Recombinant Von Willebrand Factor) Treatment Outcomes in Von Willebrand Disease in the UK: a Retrospective Chart Review Study
Brief Title: A Study on the Outcomes of Recombinant Von Willebrand Factor on Demand Treatment and Prevention and Treatment of Bleeding During and After Surgery in Adults With Inherited Von Willebrand Disease in the United Kingdom (UK)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-577-5001
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Von Willebrand Disease (VWD)
Keywords: Drug Therapy
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed With Congenital VWD: Participants who have been diagnosed with congenital VWD and prescribed rVWF within the index date range (defined as the first administration of rVWF and must fall between 1st October 2020 and 30th June 2022) will be assessed using data obtained from medical records to evaluate the treatment outcome of rVWF in real-world clinical practice.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
This study is a retrospective chart review study and will collect data on real world use of vonicog alfa (Recombinant Von Willebrand Factor [rVWF]). Von Willebrand disease (VWD) is the most common inherited bleeding disorder. rVWF is approved in Europe and UK to treat bleeding and to treat and prevent bleeding during surgeries in adults in 2018.

This study will review and collect information on the treatment and bleed prevention of adult persons with inherited VWD with rVWF in UK. These data were already collected as a part of the routine care.

The main aims of this study are to describe the use of rVWF in on-demand treatment of bleeding and the prevention of treatment and treatment of bleeding during surgeries. Other aims are to describe bleedings and their treatment as well as any surgeries before and after first treatment with rVWF and to gather information on the use of healthcare resources (such as hospital visits, emergency room visits, etc.).

ELIGIBILITY:
Inclusion criteria:

* Adults (aged 18 or over at time of first administration of rVWF) who have provided informed consent and used rVWF within its licensed indication.
* Participants who have been diagnosed with congenital von Willebrand disease.
* Confirmed instance of

  * at least one bleed (either a new bleed or ongoing bleed treated under a treatment switch) treated on-demand with rVWF between 01-Oct-2020 and 30-Jun- 2022 and/or
  * treatment to prevent and treat surgical bleeds with rVWF between 01-Oct-2020 and 30-Jun-2022

Exclusion criteria:

* Participants who were aged 17 years or less at the time of the first administration of rVWF.
* Participants who have been diagnosed with any other bleeding disorders or factor deficiencies including acquired von Willebrand disease.
* Participants with neutralising antibodies/inhibitors to VWF.
* Participants participation in a clinical trial of an investigational medical product during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been diagnosed with congenital VWD and were prescribed rVWF in UK.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Bleeding Episodes Treated with rVWF Between the Index Date and Following 12 Months | From index date up to 12 months
  Bleeding episodes will be assessed based on categories of overall and annualized, type, severity, location, bleed frequency, bleed type/location and bleed severity.
Number of Surgical Procedures Between the Index Date and Following 12 Months | From index date up to 12 months
  Surgical procedures included surgery type, severity, category (emergency or elective). Data on the participants use of rVWF in the pre-, intra- and post-operative setting during the period between the index date and the following 12 months, will be stratified by VWD type, surgery type, severity, location, or treatment rationale.
Number of Participants with Surgery Outcomes (Success, Failure, Complications) Between the Index Date and Following 12 Months | From index date up to 12 months
  Surgery outcomes (success, failure, complications) will be reported.

SECONDARY OUTCOMES:
Number of Participants With VWD-Related Healthcare Resource Utilization (HRU) | Up to 24 months
  HRU will include bleeding-related hospitalization rates, outpatient visits, accident and emergency visits.
Number of Participants With Surgery Related Costs By Type | Up to 24 months
  Surgery related costs by type will include length of stay in intensive care unit (ICU), rVWF consumption, factor VIII (FVIII) consumption, VWD treatment consumption, laboratory tests and examinations.
Number of Participants With Bleeding Episodes Treated With rVWF | Up to 24 months
  Bleeding episodes will be reported based on type, severity, location, treatment, and outcomes, of all recorded bleeds within 12 months prior to and 12 months following the first administration of rVWF.
Number of Surgical Procedures | Up to 24 months
  Surgical procedures will be reported based on surgery type (orthopaedic, gastro-intestinal, dental, etc), severity (major, minor), category (emergency or elective) treatment duration and outcomes, of all recorded surgeries within 12 months prior to and 12 months following the first administration of rVWF.
Number of Participants with Surgery Outcomes (Success, Failure, Complications) | Up to 24 months
  Surgery outcomes (success, failure, complications) based on average number of post-operative bleeds will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- United Kingdom (7):
  - University Hospitals Birmingham, Birmingham
  - Leeds Teaching Hospital, Leeds
  - Liverpool University Hospital, Liverpool
  - Royal Free London, London
  - Imperial College Healthcare, London
  - Manchester University, Manchester
  - Oxford University Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/a4acf130288f407e??page=1&idFilter=TAK-577-5001